CLINICAL TRIAL: NCT03919071
Title: A Phase 2 Study of Dabrafenib (NSC# 763760) With Trametinib (NSC# 763093) After Local Irradiation in Newly-Diagnosed BRAF V600-Mutant High-Grade Glioma (HGG)
Brief Title: Dabrafenib Combined With Trametinib After Radiation Therapy in Treating Patients With Newly-Diagnosed High-Grade Glioma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-02289; NCI-2019-02289 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS1723 (Other: Children's Oncology Group); ACNS1723 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2019-04-17; First posted 2019-04-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Astrocytoma, Not Otherwise Specified; Anaplastic Ganglioglioma; Anaplastic Pleomorphic Xanthoastrocytoma; Glioblastoma; Malignant Glioma; WHO Grade 3 Glioma; WHO Grade 4 Glioma
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Glioma | interventions — Specimen Handling; dabrafenib; Spinal Puncture; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (radiation therapy, dabrafenib, trametinib) (Experimental): Patients undergo standardized local RT 5 days a week (Monday-Friday) for 6-7 weeks. Four weeks after completion of RT, patients receive dabrafenib mesylate PO BID and trametinib dimethyl sulfoxide PO QD on days 1-28 of each cycle. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo MRI at baseline, on day 1 of cycles 1, 3, 5, 7, 11, 14, 17, 20, and 23 while on treatment, then at time of relapse, every 3 months for year 1, every 4 months for year 2, every 6 months for year 3, and annually for years 4-5. Patients may also undergo lumbar puncture for CSF testing during treatment. Patients also undergo collection of blood on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Dabrafenib Mesylate; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Drug: Trametinib Dimethyl Sulfoxide

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Dabrafenib Mesylate — Given PO
  Other Names: Dabrafenib Methanesulfonate; GSK2118436 Methane Sulfonate Salt; GSK2118436B; Tafinlar
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Trametinib Dimethyl Sulfoxide — Given PO
  Other Names: Mekinist; Meqsel; Spexotras

SUMMARY:
This phase II trial studies how well the combination of dabrafenib and trametinib works after radiation therapy in children and young adults with high grade glioma who have a genetic change called BRAF V600 mutation. Radiation therapy uses high energy rays to kill tumor cells and reduce the size of tumors. Dabrafenib and trametinib may stop the growth of tumor cells by blocking BRAF and MEK, respectively, which are enzymes that tumor cells need for their growth. Giving dabrafenib with trametinib after radiation therapy may work better than treatments used in the past in patients with newly-diagnosed BRAF V600-mutant high-grade glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the event-free survival (EFS) distribution for newly-diagnosed patients with BRAF^V600-mutant high-grade glioma (HGG) without H3 K27M mutations excluding anaplastic pleomorphic xanthoastrocytoma (aPXA) and anaplastic ganglioglioma (aGG) treated with radiation therapy followed by a maintenance combination of dabrafenib mesylate (dabrafenib) and trametinib dimethyl sulfoxide (trametinib) and to compare this EFS to contemporary historical controls.

SECONDARY OBJECTIVES:

I. To describe the overall survival (OS) distribution for newly-diagnosed patients with BRAF^V600-mutant HGG without H3 K27M mutations excluding aPXA and aGG treated with radiation therapy followed by a maintenance combination of dabrafenib and trametinib.

II. To describe the EFS and overall survival (OS) distribution for newly-diagnosed patients with BRAF^V600E-mutant aPXA and aGG without H3 K27M mutations treated with radiation therapy followed by a maintenance combination of dabrafenib and trametinib.

III. To describe the EFS and overall survival (OS) distribution for newly-diagnosed patients with BRAF^V600E-mutant HGG including aPXA and aGG with H3 K27M mutations treated with radiation therapy followed by a maintenance combination of dabrafenib and trametinib.

IV. To define and evaluate the toxicities of combination therapy with dabrafenib and trametinib after radiation therapy in newly-diagnosed patients with HGG.

EXPLORATORY OBJECTIVE:

I. To bank tumor specimens and body fluids (blood, urine and cerebrospinal fluid) for future studies.

OUTLINE:

Patients undergo standardized local radiation therapy (RT) 5 days a week (Monday-Friday) for 6-7 weeks. Four weeks after completion of RT, patients receive dabrafenib mesylate orally (PO) twice daily (BID) and trametinib dimethyl sulfoxide PO once daily (QD) on days 1-28 of each cycle. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a magnetic resonance imaging (MRI) at baseline, on day 1 of cycles 1, 3, 5, 7, 11, 14, 17, 20, and 23 while on treatment, then at time of relapse, every 3 months for year 1, every 4 months for year 3, every 6 months for year 3, and annually for years 4-5. Patients may also undergo lumbar puncture for cerebral spinal fluid (CSF) testing during treatment. Patients also undergo collection of blood on study.

After completion of study treatment, patients are followed up at disease relapse, every 3 months for year 1, every 4 months for year 2, every 6 months for year 3, then annually for years 4-5.

ELIGIBILITY:
Inclusion Criteria:

* PRE-ENROLLMENT ELIGIBILITY SCREENING: Patients must be =< 25 years of age at the time of enrollment on APEC14B1 Part A CNS/HGG pre-enrollment eligibility screening.

  * Note: This required age range applies to the pre-enrollment eligibility screening for all HGG patients. Individual treatment protocols may have different age criteria.
* PRE-ENROLLMENT ELIGIBILITY SCREENING: Patient is suspected of having localized newly-diagnosed HGG, excluding metastatic disease.
* PRE-ENROLLMENT ELIGIBILITY SCREENING: Patient and/or their parents or legal guardians have signed informed consent for eligibility screening on APEC14B1 Part A.
* PRE-ENROLLMENT ELIGIBILITY SCREENING: The specimens obtained at the time of diagnostic biopsy or surgery must be submitted through APEC14B1 as soon as possible (ASAP), preferably within 5 calendar days of the procedure.

  * Please note: See the APEC14B1 Manual of Procedures for a full list of detailed instructions for submitting required materials and for shipping details.
* Patients must be >= 3 years and =< 25 years of age at the time of enrollment.
* Patients must have eligibility confirmed by Rapid Central Pathology and Molecular Screening Reviews performed on APEC14B1:

  * Newly diagnosed high-grade glioma with BRAF^V600-mutation
  * Results for H3 K27M by immunohistochemistry (IHC) or sequencing
  * Histologically confirmed high-grade glioma (World Health Organization [WHO] grade III or IV) including but not limited to: anaplastic astrocytoma (AA), anaplastic pleomorphic xanthoastrocytoma (aPXA), anaplastic gangliogliomas (aGG), glioblastoma (GB), and high-grade astrocytoma, not otherwise specified (NOS).
* Patients must have had histologic verification of a high-grade glioma diagnosis. CSF cytology by lumbar puncture must be done if clinically indicated and determined to be safe prior to study enrollment. If cytology proves positive, the patient would be considered to have metastatic disease and would, therefore, be ineligible.
* A pre- and post-operative brain MRI with and without contrast and a baseline spine MRI with contrast must be obtained prior to enrollment. The requirement for a post-operative MRI is waived for patients who undergo biopsy only. If the spine MRI is positive, the patient would be considered to have metastatic disease and would be ineligible.
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age.
* Peripheral absolute neutrophil count (ANC) >= 1000/uL (within 7 days prior to enrollment).
* Platelet count >= 100,000/uL (transfusion independent) (within 7 days prior to enrollment).
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions) (within 7 days prior to enrollment).
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 (within 7 days prior to enrollment) or
* A serum creatinine based on age/sex as follows (within 7 days prior to enrollment):

  * Age 3 to < 6 years (Male 0.8 mg/dL, Female 0.8 mg/dL)
  * Age 6 to < 10 years (Male 1 mg/dL, Female 1 mg/dL)
  * Age 10 to < 13 years (Male 1.2 mg/dL, Female 1.2 mg/dL)
  * Age 13 to < 16 years (Male 1.5 mg/dL, Female 1.4 mg/dL)
  * Age >= 16 years (Male 1.7 mg/dL, Female 1.4 mg/dL)

    * The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the Centers for Disease Control and Prevention (CDC).
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment), and
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (within 7 days prior to enrollment). For the purpose of this study, the ULN for SGPT is 45 U/L.
* Patients with a seizure disorder may be enrolled if their seizures are well controlled while on non-enzyme inducing anticonvulsants permitted on this study.
* Patients must be enrolled and protocol therapy must be projected to begin no later than 31 days after definitive surgery (day 0). If a biopsy only was performed, the biopsy date will be considered the date of definitive surgery. For patients who have a biopsy or incomplete resection at diagnosis followed by additional surgery, the date of the last resection will be considered the date of definitive surgery.
* All patients and/or their parents or legal guardians must sign a written informed consent.

Exclusion Criteria:

* Patients with intrinsic brainstem or primary spinal cord tumors will be excluded.
* Patients with metastatic disease (defined as neuraxis dissemination either by imaging or by cytology) will be excluded.
* Patients must not have received any prior tumor-directed therapy including chemotherapy, radiation therapy, immunotherapy, or bone marrow transplant for the treatment of HGG other than surgical intervention and/or corticosteroids.
* Previous treatment with dabrafenib or another RAF inhibitor, trametinib or another MEK inhibitor, or an ERK inhibitor.
* Patients with a history of a malignancy with confirmed activating RAS mutation.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dabrafenib, trametinib, and their excipients.
* Uncontrolled medical conditions (e.g., diabetes mellitus, hypertension, liver disease, or uncontrolled infection), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol.
* Presence of active gastrointestinal (GI) disease or other condition (e.g., small bowel or large bowel resection) that will interfere significantly with the absorption of drugs.
* History of hepatitis B virus, or hepatitis C virus infection (patients with laboratory evidence of cleared hepatitis B virus and/or hepatitis C virus may be enrolled).
* History or current diagnosis of cardiac disease indicating significant risk of safety for patients participating in the study such as uncontrolled or significant cardiac disease, including any of the following:

  * Recent myocardial infarction (within the last 6 months);
  * Uncontrolled congestive heart failure;
  * Unstable angina (within last 6 months);
  * Clinically significant (symptomatic) or known, uncontrolled cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third degree atrioventricular [AV] block without a pacemaker) except sinus arrhythmia within the past 24 weeks prior to the first dose of study treatment;
  * Coronary angioplasty or stenting (within last 6 months);
  * Intra-cardiac defibrillators;
  * Abnormal cardiac valve morphology (>= grade 2) documented by echocardiogram.
* Patients with a history or current evidence of retinal vein occlusion (RVO) or central serous retinopathy (CSR), or predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension).
* Patients with presence of interstitial lung disease or pneumonitis.
* Female patients who are pregnant are ineligible since there is yet no available information regarding human fetal or teratogenic toxicities.
* Lactating females are not eligible unless they have agreed not to breastfeed their infants for the duration of the study and for 4 months following discontinuation of study therapy.
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained.
* Sexually active patients of reproductive potential (male or female) are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation and for 4 months following discontinuation of study therapy. Male patients (including those who have had a vasectomy) taking dabrafenib and trametinib combination therapy must use a condom during intercourse while on study and for 16 weeks after stopping treatment, and should not father a child during these periods. Women of childbearing potential should use effective non-hormonal contraception during therapy and for 4 weeks following discontinuation of dabrafenib and at least 4 months following the last dose of trametinib in patients taking combination therapy. Women should be advised that dabrafenib may decrease the efficacy of hormonal contraceptives and an alternate method of contraception, such as barrier methods, should be used.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) for stratum 1 | From the date of diagnosis until disease progression date, secondary malignant neoplasm occurrence date, death date of any cause, or last follow-up, assessed up to 5 years
  The EFS curve for the new treatment cohort (stratum 1) will be estimated by Kaplan Meier estimates. A 2-sample, 1 sided log-rank test will be used to test whether the EFS distribution is better in new treatment compared with historical control. Calculation of the EFS will be based on the site determination as central review will be performed retrospectively.

SECONDARY OUTCOMES:
Overall survival (OS) for stratum 1, stratum 2, and stratum 3 | From the date of diagnosis until death date of any cause or last follow up date, assessed up to 5 years
  The OS curve for the new treatment cohort (stratum 1) will be estimated by Kaplan Meier estimates. A 2-sample, 1 sided log-rank test will be used to test whether the OS distribution is better in new treatment compared with historical control. For stratum 2 and stratum 3, Kaplan Meier estimates will be provided for OS distribution.
Event-free survival (EFS) for stratum 2 and stratum 3 | Follow up date, assessed up to 5 years
  For stratum 2 and stratum 3, Kaplan Meier estimates will be provided for EFS distribution.
Incidence of adverse events | Up to 5 years
  Graded per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Grade 3 and higher toxicities observed by cycle will be listed for each stratum separately. The grade 3 and higher toxicities observed by cycle and by system organ class for the eligible patients will also be listed for each stratum separately. Toxicity data will be reported separately for the radiation therapy phase versus the maintenance therapy phase for clarity of attribution. Toxicity monitoring will include toxicities such as grade 2 or higher pyrexia, uveitis, retinal vein occlusion, retinal pigment epithelial detachment, and decreased left ventricular ejection fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Rishi R Lulla, Principal Investigator — Children's Oncology Group
Locations (131):
- United States (130):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Shahid S, Kushner BH, Modak S, Basu EM, Rubin EM, Gundem G, Papaemmanuil E, Roberts SS. Association of BRAF V600E mutations with vasoactive intestinal peptide syndrome in MYCN-amplified neuroblastoma. Pediatr Blood Cancer. 2021 Oct;68(10):e29265. doi: 10.1002/pbc.29265. Epub 2021 Jul 31. PMID 34331515

DOCUMENTS (1):
  • Informed Consent Form (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT03919071/ICF_000.pdf